CLINICAL TRIAL: NCT00969800
Title: Double-blind Sham Device-controlled Multi-center Crossover Trial of Chlorine Dioxide Gas on the Protective Effect Against Respiratory Infections
Brief Title: Test of a Preventive Effect of a Deodorant Device Against Respiratory Infections
Acronym: Cleverin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taiko Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Norio Ogata, MD, PhD, Taiko Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: TA90811
Record Dates: First submitted 2009-08-30; First posted 2009-09-01 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Respiratory Infection
Keywords: Common cold; Influenza; Pneumonia
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Influenza, Human; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Cleverin Gel (Experimental): Active Cleverin Gel, which generates chlorine dioxide gas, is placed in a room of subject.
  Interventions: Device: Cleverin Gel
- Inactive Cleverin Gel (Sham Comparator): Inactive Cleverin Gel is placed in a room of subject. It does not generate chlorine dioxide gas.
  Interventions: Device: Inactive Cleverin Gel

INTERVENTIONS:
Device: Cleverin Gel — Chlorine dioxide gas concentration at a range of 0.005 to 0.03 ppm.
  Other Names: ClO2 gas generator
  Arms: Active Cleverin Gel
Device: Inactive Cleverin Gel — Seemingly same chlorine dioxide gas-generating device, but no gas is generated.
  Other Names: sham ClO2 gas generator
  Arms: Inactive Cleverin Gel

SUMMARY:
This study is to test whether a chlorine dioxide gas-generating device, which releases a low concentration gas of chlorine dioxide in a sustained manner, can protect against respiratory infections in elderly individuals living in nursing homes. Such a device is used as a deodorant for normal domestic purposes. The investigators reasoned that the antiviral and antibacterial properties of chlorine dioxide might lead to a lowering in the incidence of respiratory infectious diseases. The study is designed as a randomized placebo-controlled double-blind crossover multicentre trial involving approximately 1500 subjects.

DETAILED DESCRIPTION:
Chlorine dioxide (ClO2), which is used as household deodorant, is a volatile gas that displays very strong oxidative activity. Indeed, the powerful oxidative activity of chlorine dioxide (Ogata, N., Biochemistry 46, 4898-4911, 2007) is responsible for its antimicrobial activity against bacteria (Benarde, M. A., et al. Appl. Mircrobiol. 15, 257-265, 1967), fungi (Morino, H., et al. Yakugaku Zasshi 127, 773-777, 2007) and viruses (Ogata, N. and Shibata, T. J. Gen. Virol. 89, 60-67, 2008). Recently, we found that the rate of absenteeism due to illness in a school was lower in classrooms where a chlorine dioxide gas-generating device was placed than in classrooms with no such device. Based upon this unexpected observation we hypothesize that chlorine dioxide gas, at a concentration low enough not to harm humans, may lower the incidence of respiratory infections by inactivating airborne microorganism within an enclosed space.

ELIGIBILITY:
Inclusion Criteria:

* Those who who agrees with the aim of the study

Exclusion Criteria:

* Those who do not agree with the aim of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1469 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The number of incidence of respiratory infections | Four months

SECONDARY OUTCOMES:
The incidence of adverse effects | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Norio Ogata, MD, PhD, Principal Investigator — Taiko Pharmaceutical Co., Ltd.
Locations (1):
- Reifuen Nursing Home, Osaka, Osaka, Japan